CLINICAL TRIAL: NCT03447509
Title: Grasping Function After Spinal Cord Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: funding ended
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: B2474-R
Record Dates: First submitted 2018-01-31; First posted 2018-02-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injury
Keywords: Spinal cord injury; neural control; motor function; hand movement
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Magnetic Stimulation and Acoustic Startle
Who Masked: Participant
Masking Description: Participants will not know if they receive real or sham Stimulation and/or real or sham Startle
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experiment 1a (Active Comparator): Examine physiological mechanisms contributing to the control of precision and power grip behaviors. To accomplish this aim the investigators propose to complete one main experiment. The investigators will test the hypotheses that there are two fundamentally distinct modes of hand operation after SCI. One involves brainstem pathways, and permits whole-hand 'power grip', while the other involves corticospinal and motor cortical connections, and allows a wide range of fractionated finger movements (precision grip) after SCI. Measurements of corticospinal, reticulospinal, and motoneuron excitability will be tested during index finger abduction, precision and power grip.
  Interventions: Device: iTMS; Other: Motor Task
- Experiment 1b (Active Comparator): To accomplish this aim the investigators propose to complete one main experiment. The investigators will use iTMS and/or an acoustic startle stimuli to test the hypothesis that induced-plasticity protocols (iTMS and startle stimuli) will enhance EMG and force output in hand muscles during grasping. In a randomized sham crossover design, SCI and controls will be assigned to two groups: (1) iTMS applied during precision and power grip (two randomized sessions), and (2) startle applied during precision and power grip (two randomized sessions).
  Interventions: Device: iTMS; Other: Motor Task
- Experiment 2 (Active Comparator): To accomplish this aim the investigators propose to complete one main experiment. The investigators will combine iTMS and/or acoustic startle with precision and power grip training to test the hypothesis that 'precision and power grip training outcomes will be enhanced by iTMS and startle induced plasticity'. In a randomized sham controlled design, SCI and control subjects will be assigned to: training+iTMS and training+sham iTMS and training+startle and training+sham startle.
  Interventions: Device: iTMS; Other: Motor Task; Device: Sham iTMS; Other: Training

INTERVENTIONS:
Device: iTMS — Small magnetic pulse will be given to the brain in a non invasive manner.
Other: Motor Task — Participants will be asked to perform specific motor tasks or movements with their fingers, hands, and arms.
Device: Sham iTMS — Sham or fake stimulation will be given to the brain in a non invasive manner.
  Arms: Experiment 2
Other: Training — The participant will be instructed to do repetitive motor movements with their arm or hand.
  Arms: Experiment 2

SUMMARY:
The overall goals of this proposal are to examine the contribution of physiological pathways to the control of grasping behaviors after cervical SCI, and to maximize the recovery of grasping by using tailored non-invasive brain stimulation and acoustic startle protocols with motor training. The investigators propose to study two basic grasping behaviors, which are largely used in most daily-life activities: a precision grip and a power grip.

DETAILED DESCRIPTION:
Grasping behaviors, which are essential for daily-life functions, are largely impaired in individuals with cervical spinal cord injury (SCI). Although rehabilitative interventions have shown success in improving the ability to grasp following injury their overall effects remain limited. The goals of this proposal are to examine the contribution of physiological pathways to the control of grasping behaviors after cervical SCI, and to maximize the recovery of grasping by using tailored non-invasive stimulation protocols with motor training. The investigators propose to study two basic grasping behaviors: a precision grip and a power grip. These behaviors are crucial because they provide the basis for a number human prehensile manipulations and are also necessary skills for eating, writing, dressing, and many other functions. Thus, the study results may have a direct impact on the quality of life for Veterans and their caregivers by enhancing their independence and level of care.

In Aim 1, the investigators will investigate the contribution of corticospinal and brainstem pathways to the control of hand muscles involved in precision and power grip after cervical SCI. Transcranial magnetic stimulation (TMS) will be used to examine transmission in corticospinal and intracortical pathways targeting finger muscles and an acoustic startle stimulus with and without TMS will be used to examine the contribution from brainstem pathways.

In Aim 2, the investigators propose to enhance the recovery of grasping by using novel tailored protocols of non-invasive repetitive TMS targeting late indirect (I) descending volleys (iTMS) and an acoustic startle stimuli. iTMS and startle will be used during precision and power grip movements in a task-dependent manner to induce cortical and subcortical plasticity and enhance voluntary output of hand muscles. Later, iTMS and startle will be applied in a task-dependent manner during a motor training task that involves precision and power grip. These unique approaches aim at promoting neuroplasticity during functionally relevant grasping movements has not been used before.

ELIGIBILITY:
Inclusion Criteria:

Participants who are unimpaired healthy controls:

* Male and females between ages 18-85 years
* Right handed
* Able to complete precision grips with both hands
* Able to complete full wrist flexion-extension bilaterally

Participants who have had a spinal cord injury:

* Male and females between ages 18-85 years
* Chronic SCI (> 1 year post injury)
* Spinal Cord injury at C8 or above
* Intact or impaired but not absent innervations in dermatomes C6. C7 and C8 during light touch and pin prick stimulus using the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) sensory scores
* The ability to produce a visible precision grip force with one hand
* Able to perform some small wrist flexion and extension
* ASIA A,B,C, or D

Exclusion Criteria:

Exclusion criteria for enrollment For SCI and Healthy Control Subjects (4-8 exclusion for non-invasive brain stimulation only):

* Uncontrolled medical problems including pulmonary, cardiovascular or orthopedic disease
* Any debilitating disease prior to the SCI that caused exercise intolerance
* Premorbid, ongoing major depression or psychosis, altered cognitive status
* History of head injury or stroke
* Pacemaker
* Metal plate in skull
* History of seizures
* Receiving drugs acting primarily on the central nervous system, which lower the seizure threshold
* Pregnant females
* Ongoing cord compression or a syrinx in the spinal cord or who suffer from a spinal cord disease such as spinal stenosis, spina bifida, MS, or herniated disk

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in amplitude of Motor evoked potential size | Post treatment at minute 0, minute 10, minute30, minute 60.
  At the stated minute interval TMS measurements are reassessed.

SECONDARY OUTCOMES:
Grip Strength and 9-hole peg test | Post treatment at minute 0, minute 10, minute30, minute 60.
  At the stated minute interval the following measurements are reassessed: Force is measured during a grip task as muscle electrical activity (electromyography) is recorded in millivolts (mV) and 9-hole peg test is a dexterity measure, estimated as the time required to complete the task (seconds).

CONTACTS AND LOCATIONS:
Overall Officials: Monica A Perez, PhD, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (1):
- Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-08-29): https://cdn.clinicaltrials.gov/large-docs/09/NCT03447509/ICF_000.pdf